CLINICAL TRIAL: NCT06981949
Title: The Addition of Dexmedetomidine to Ropivacaine in Bilateral Erector Spinae Plane Block in Patients Undergoing Coronary Artery Bypass Surgery - A Double-blinded Randomized Clinical Trial
Brief Title: Addition of Dexmedetomidine to Ropivacaine in Bilateral Erector Spinae Plane Block in Patients Undergoing Coronary Artery Bypass Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Lebanese American University (Other)
Responsible Party: Principal Investigator, Caroline Chahine, Clinical Instructor of Medicine, Lebanese American University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAUMCRH.CC1.23/Apr/2025
Record Dates: First submitted 2025-05-03; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Pain; Pain Management Following Cardiopulmonary Bypass Surgery; Erector Spinae Plane Block
MeSH Terms: conditions — Pain | interventions — Dexmedetomidine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group Ropivacaine Only (R) (Active Comparator): In Group R, patients will receive 20 ml of 0.375% ropivacaine in each side of a bilateral single-shot ultrasound-guided erector spinae plane block.
  Interventions: Drug: Ropivacaine
- Group Combination Ropivacaine and Dexmedetomidine (RD) (Experimental): In Group RD, patients will receive 20 ml of 0.375% ropivacaine plus 0.5 micrograms/kg of dexmedetomidine in each side of a bilateral single-shot ultrasound-guided erector spinae plane block.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine added to ropivacaine in the bilateral single-shot Ultrasound-guided erector spinae plane block that will be applied to each side (bilateral):
  20ml/side of 0.375% ropivacaine+0.5 μg/kg/side of dexmedetomidine (lean body weight if BMI >30)
  Arms: Group Combination Ropivacaine and Dexmedetomidine (RD)
Drug: Ropivacaine — Ropivacaine only in the Bilateral single-shot Ultrasound-guided Erector Spinae Plane Block:
  20ml/side of 0.375% ropivacaine
  Arms: Group Ropivacaine Only (R)

SUMMARY:
Coronary artery bypass surgery (CABG), typically performed through a median sternotomy, causes significant postoperative pain. Managing this pain effectively while reducing reliance on opioids is essential, as opioids can lead to side effects such as respiratory depression, nausea, and potential for dependence. Regional anesthesia techniques like the erector spinae plane block (ESPB) have emerged as promising tools to control pain and support recovery.

This randomized, double-blind clinical trial evaluates whether adding dexmedetomidine, a sedative and analgesic, to ropivacaine, a local anesthetic, in bilateral ESPB can improve pain control after off-pump CABG surgery. The study is conducted at the Lebanese American University Medical Center - Rizk Hospital.

A total of 110 adult patients undergoing elective surgery are randomly assigned to one of two groups:

1. Group R: Receives ropivacaine alone in the ESPB.
2. Group RD: Receives ropivacaine with dexmedetomidine.

The nerve block is administered before anesthesia. The primary outcome is the duration of effective pain relief (pain score ≤4) before the patient needs opioid medication, assessed up to 24 hours after extubation.

Secondary outcomes include:

1. Pain scores monitored for up to 48 hours post-extubation
2. Total intraoperative opioid use
3. Time to extubation, ambulation, and incentive spirometry use
4. ICU stay duration
5. Side effects such as nausea, bradycardia, or local anesthetic toxicity

This study supports efforts to reduce opioid use after heart surgery while maintaining effective pain management, aligning with enhanced recovery protocols and addressing the broader public health challenge of opioid overuse.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 25 - 80 years old
2. Planned for elective OFF PUMP CABG
3. Cognitively not impaired
4. American Society of Anesthesiologists class 3
5. Left ventricular ejection fraction ≥40%
6. Consent form for the study signed
7. No infection at the site of injection
8. No contraindication for ESP block (thrombocytopenia, anticoagulation therapy)
9. No documented allergy to ropivacaine or dexmedetomidine

Exclusion Criteria:

1. Refusal to participate in the study
2. Emergency surgery
3. American Society of Anesthesiologists class >3
4. Left ventricular ejection fraction <40%
5. Infection at the site of injection for ultrasound-guided ESPB
6. Coagulation disorders
7. Documented allergy to ropivacaine or dexmedetomidine
8. Greater than first-degree heart block
9. Bradycardia (heart rate [HR] < 50 bpm)
10. Pregnancy
11. BMI ≥40
12. Psychiatric illnesses that would interfere with the assessment of pain scores
13. History of alcohol or drug abuse and chronic analgesic use

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-16 (Estimated)

PRIMARY OUTCOMES:
Analgesia time | From the moment the patient is awake in the Intensive Care Unit until the end of the patient's study inclusion time (48 hours after extubation)
  The period during which the pain numerical rating scale score remains less than or equal to 4 and until the time the patient required the administration of opioid as the first administration. The numerical rating scale score is a 0-10 scale, where 0 represents "no pain" and 10 represents "worst pain imaginable".

SECONDARY OUTCOMES:
Total intraoperative opioid | Intraoperatively
  Total intraoperative opioid usage in terms of morphine equivalent
Total amount of rescue analgesics used | Postoperatively until 48 hours post-extubation
  Rescue analgesia requirements, including morphine or other than morphine, includes the total amount of each rescue analgesic used
Pain score | Postoperatively until 48 hours post-extubation
  Pain scores postoperatively related to chest pain: measured using the numerical rating scale to get pain scores on pre-specified time points. The minimum score is 0, "no pain at all," and the maximum score is 10, "worst possible pain."

OTHER OUTCOMES:
Time to extubation | Perioperative
Time to first incentive spirometry use | Perioperative
Time to ambulation | Perioperative
Total length of ICU stay | Perioperative
Sedation score | Perioperative
  Sedation score postextubation measured using the Ramsay Sedation Scale. The Ramsay Sedation Scale ranges from 1 to 6, where 1 signifies "Awake; agitate or restless or both" and 6 signifies "asleep; no response to glabellar tap or loud auditory stimulus".

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified research-related clinical data will be shared on reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: After the publication of the study manuscript.
Access Criteria: Researchers will be able to access the IPD and supporting information mentioned above only with a reasonable request. After assessment and in the case of approval, a data sharing agreement must be made between the study PI, the study institutional review board, and the researcher/entity requesting the de-identified dataset.